CLINICAL TRIAL: NCT00414635
Title: A Randomized Controlled Trial of a Weekly Schedule of Five Consecutive Days on Treatment With Efavirenz, Tenofovir, and Emtricitabine Followed by Two Days Off Treatment (5/2 Intermittent Treatment Schedule) Versus Continuous Treatment in Individuals With Virologic Suppression on This Combination
Brief Title: FOTO: Five Consecutive Days on Treatment With Efavirenz, Tenofovir, and Emtricitabine Followed by Two Days Off Treatment Versus Continuous Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Collaborators: The Campbell Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-156
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; efavirenz; tenofovir; emtricitabine; FOTO; treatment interruption; Atripla; Truvada; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This study is designed to compare the control and the experimental arm groups for 24 weeks of treatment. After 24 weeks, subjects on the control arm then cross over to the experimental intervention.

ARMS (2):
- Control Arm with Week 24 Crossover (Other): Subjects randomized to the control arm will remain on daily dosing of the pre-study regimen of 600mg efavirenz and 1 coformulated tablet of 300mg tenofovir df + 200 mg emtricitabine by mouth daily, or the equivalent coformulated single tablet of 600mg efavirenz + 300mg tenofovir df + 200 mg emtricitabine by mouth daily for 24 weeks. After 24 weeks of daily therapy subjects on this arm may be eligible to cross over to the experimental arm regimen of the coformulated single tablet of 600 mg efavirenz +300 mg tenofovir df +200 mg of emtricitabine on the 5/2 intermittent dosing treatment schedule for the remainder of the study.
  Interventions: Drug: Intermitent Dosing
- 5/2 Intermitent Treatment Arm (Experimental): Subjects randomized to the 5/2 intermittent dosing treatment schedule regimen will be prescribed the pre-study regimen of 600mg efavirenz and 1 coformulated tablet of 300mg tenofovir df + 200 mg emtricitabine by mouth daily, or the equivalent coformulated single tablet of 600mg efavirenz + 300mg tenofovir df + 200 mg emtricitabine by mouth daily, for 5 consecutive days per week followed by 2 days off of these medications, 600 mg efavirenz, 300 mg tenoforvir dt and 200 mg emtricitabine, for 48 weeks.
  Interventions: Drug: Intermitent Dosing

INTERVENTIONS:
Drug: Intermitent Dosing — Intermittent dosing treatment is the maintenance of the "5/2" schedule, where the regimen, 300 mg tenofovir td, 600 mg efavirenz, 200 mg emtricitabine is dosed for 5 consecutive days - typically Monday through Friday - followed by two days off of medication, 300 mg tenofovir td, 600 mg efavirenz, 200 mg emtricitabine. .

SUMMARY:
For people with HIV who are currently taking specific medications (including Sustiva (efavirenz)) and have no detectable viral load, this study tracks how patients do if they take their medications for five days of the week compared with seven days of the week.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate virologic control of a weekly schedule of 5 days of treatment followed by two days off treatment versus continuous treatment with the same regimen. This is a larger study based on the results of our successful pilot study using the same protocol. The 48 week, phase IV trial addresses the issues of the high cost of HIV treatment, adherence problems associated with daily treatment, and cumulative toxicities. Virologic and immunologic parameters, drug levels of efavirenz, adherence, and toxicity will be measured. Subjects will have to be seen at CRI for 6 visits after randomization. Subjects randomized to daily therapy will cross over to 5/2 therapy at 24 weeks if their viral load remains undetectable.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* CD4 count > or = 200
* Viral load < 50
* Treatment with a regimen containing efavirenz and tenofovir and lamivudine or emtricitabine for at least 90 days prior to screening

Exclusion Criteria:

* Detectable HIV RNA on an ultrasensitive assay within the 90 days preceding screening
* Prior evidence of intermediate or high level resistance to efavirenz, tenofovir or cytidine analogues
* Hepatitis B infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin J Cohen, MD, MSc, Principal Investigator — CRI
Locations (7):
- United States (7):
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - CARE-ID, Washington D.C., District of Columbia
  - Steinhart Medical Associates, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Treasure Chest Infectious Disease, Vero Beach, Florida
  - Community Research Initiative of New England - Boston, Boston, Massachusetts
  - Community Research Initiative of New England - West, Springfield, Massachusetts

REFERENCES:
- See also: Web page of CRI, the nonprofit research group sponsoring the study — http://www.crine.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between August 21, 2006 and November 9, 2007. Recruitment occured at multiple site locations (research clinics and private practice).
Groups:
- FOTO: Participants changing to 5 days on, 2 days off (FOTO). The 5/2 intermittent treatment arm will take their antiretrovirals for 5 consecutive days followed by 2 days off for 48 weeks (provided their HIV RNA remains undetectable on an ultrasensitive assay).
- Control: Daily regimen (7 days)• The control arm will take their antiretrovirals for 7 days a week for the first 24 weeks and then cross over to the 5/2 intermittent treatment schedule (if their HIV RNA remains undetectable on an ultrasensitive assay) for the remainder of the study.
Period: Overall Study
Arm/Group | FOTO | Control
Started | 30 | 30
Completed | 25 | 28
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOTO | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 28 | 58
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.1) | 47 (9.9) | 44 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Virologic Suppression (Less Than 50 RNA Cps/ml)
Description: Percentage of Participants maintaining full Virologic Suppression (less than 50 RNA cps/ml)
Time Frame: 24 weeks
Population: Per protocol
Measure: Number; unit: Percentage of Participants
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 28
Percentage of Participants | 100 | 86

2. Secondary Outcome: Mean CD4+ T-cell Count Increases From Baseline to Week 24.
Time Frame: Baseline to Week 24
Measure: Mean (95% Confidence Interval); unit: cells/ml
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 28
cells/ml | -1.9 [-50.6 to 46.9] | -9.3 [-57.9 to 39.3]

3. Secondary Outcome: Quality of Life
Description: Participant preference of antiretroviral (ART) regimen determined on a scale ranging from 0 to 10. O was defined as "I Perfer taking HIV medications 7 days/week" and 10 was defined as "I perfer 5 days on and 2 days off". We present results of a single question on quality of life experienced while on their study ART regimen.
Time Frame: 4 weeks
Population: The questionnaire was only applicable to FOTO arm
Measure: Median (Inter-Quartile Range); unit: Units on a Scale
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 0
Units on a Scale | 9.5 [8 to 10] |

4. Secondary Outcome: Absolute Number of Virological "Blip" Events Occurring Over 24 Weeks
Description: Total number of "blip" events in each arm. Blips are defined as HIV RNA > 50 and < 200 cps/ml
Time Frame: Baseline to week 24
Measure: Number; unit: blip events
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 28
blip events | 8 | 10

5. Secondary Outcome: Trough Blood Levels of Efavirenz in Both Arms
Description: blood levels of efavirenz measured at 60 hours post last dose in FOTO arm and 12 hours post last dose in daily arm (control)
Time Frame: 12 or 60 hours
Measure: Number; unit: Percentage of Participants
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 28
Percentage of Participants
  >1000 nanograms/milliliter (ng/ml) | 48 | 90
  500-999 nanograms/milliliter (ng/ml) | 37 | 1
  <500 nanograms/milliliter (ng/ml) | 15 | 9

6. Secondary Outcome: Self-reported Adherence Summary in Both Arms
Description: Percentage of participants who missed one or more doses in weekly regimen.
Time Frame: 4, 12 and 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 28
percentage of participants
  Week 4 | 10 | 17
  Week 12 | 15 | 7
  Week 24 | 8 | 11

7. Secondary Outcome: Deviation From FOTO Schedule by One Extra Dose
Description: Percentage of FOTO participants who took a dose during weekend planned interuption period
Time Frame: 4, 12, 24 weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | FOTO | Control
Number analyzed (Participants) | 25 | 0
Percentage of Participants
  Week 4 | 10 |
  Week 12 | 4 |
  Week 24 | 8 |

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | FOTO | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/30
Other Adverse Events (participants affected / at risk) | 6/30 | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOTO (N=30) | Control (N=30)
melonoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hospitalization status post cardiac catherization (General disorders) | 0 (0) | 1 (1)
hospitalization status post gastric banding procedure (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOTO (N=30) | Control (N=30)
Cough (General disorders) | 2 (2) | 5 (5)
nightsweats (General disorders) | 0 (0) | 3 (3)
sinusitis (General disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
Conclusions are limited by the small "n" studied. The results are only applicable to the specific drug regimen studied and thus can not be generalized to all ART. We only studied individuals already virologically undetectable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site investigators agree not to individually publish the results of the study. They may participate in a joint publication of the study results with the sponsor.